CLINICAL TRIAL: NCT03030209
Title: Risk Factors for the Development of Diabetes Mellitus After Distal Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-GS03
Record Dates: First submitted 2016-09-17; First posted 2017-01-24 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
Keywords: pancreatectomy; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Distal Pancreatectomy: Patients undergoing distal pancreatectomy
  Interventions: Procedure: Distal pancreatectomy

INTERVENTIONS:
Procedure: Distal pancreatectomy — Distal pancreatectomy with or without splenectomy using minimal invasive or open approach

SUMMARY:
Glucose homeostasis changes after distal pancreatectomy are not well understood. This study aim to identify the incidence of and risk factors for, a change in glucose homeostasis in patients who underwent distal pancreatic resection.

DETAILED DESCRIPTION:
The development of sophisticated surgical procedures, improved postoperative care, and the capacity for early diagnosis of disease, have prolonged life expectancy after pancreatic resection. For these patients, the endocrine function of the pancreas is a critical factor that influences quality of life. In this study, the investigators recruit patients who underwent distal pancreatectomy in Peking Union Medical College Hospital within the last 10 years. Demographic characteristics, operative parameters and short-term postoperative outcomes were collected in a prospective database maintained by the Pancreatic Surgical Centre, Peking Union Medical College Hospital. These patients are followed up regularly by outpatient visiting or telephone for long-term outcomes. The primary outcome of this study is new-onset diabetes mellitus; second outcomes include impaired fasting glucose, impaired glucose tolerance, exocrine insufficiency and disease recurrence. This study aim to determine the cumulative rates of endocrine insufficiency, and identify risk factors for DM development in a large cohort of patients undergoing distal pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing distal pancreatectomy

Exclusion Criteria:

* Patients undergoing pancreaticoduodenectomy, middle pancreatectomy and enucleation
* Patients with preoperative DM
* Patients with functioning insulinoma and multiple endocrine neoplasia type 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing distal pancreatectomy at our single tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2016-02-13 (Actual); Study Completion 2016-02-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with new-onset diabetes mellitus as defined by American Diabetes Association | Through study completion, an average of 3 year
  The criteria for the diagnosis of diabetes developed by American Diabetes Association (1) FPG (fasting plasma glucose) ≥ 126 mg/dL (7.0 mmol/L). Fasting is defined as no caloric intake for at least 8 h.* OR (2) 2-h PG (plasma glucose) ≥ 200 mg/dL (11.1mmol/L) during an OGTT (oral glucose tolerance test). The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water.* OR (3) A1C ≥ 6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is NGSP certified and standardized to the DCCT assay.* (lower-upper limit: 4.5%-6.3% in PUMCH) OR (4) In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥ 200 mg/dL (11.1 mmol/L).
  *In the absence of unequivocal hyperglycemia, results should be confirmed by repeat testing.

SECONDARY OUTCOMES:
Number of participants with new-onset prediabetes as defined by American Diabetes Association | Through study completion, an average of 3 year
  The categories of prediabetes (increased risk for diabetes)
  (1) Impaired fasting glucose (IFG): FPG 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L). (3.6 - 6.1 mmol/L in PUMCH) OR (2) Impaired glucose tolerance (IGT): 2-h PG in the 75-g OGTT 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L). The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water.
  OR (3) A1C 5.7-6.4% (39-46 mmol/mol)
Number of participants with new-onset exocrine insufficiency | Through study completion, an average of 3 year
  Exocrine insufficiency is defined as patients requiring oral pancreatic enzyme replacement because of severe diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, M.D., Study Chair — Department of General Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwon JH, Kim SC, Shim IK, Song KB, Lee JH, Hwang DW, Park KM, Lee YJ. Factors Affecting the Development of Diabetes Mellitus After Pancreatic Resection. Pancreas. 2015 Nov;44(8):1296-303. doi: 10.1097/MPA.0000000000000404. PMID 26390413
- [Background] Shirakawa S, Matsumoto I, Toyama H, Shinzeki M, Ajiki T, Fukumoto T, Ku Y. Pancreatic volumetric assessment as a predictor of new-onset diabetes following distal pancreatectomy. J Gastrointest Surg. 2012 Dec;16(12):2212-9. doi: 10.1007/s11605-012-2039-7. Epub 2012 Sep 28. PMID 23054900
- [Background] King J, Kazanjian K, Matsumoto J, Reber HA, Yeh MW, Hines OJ, Eibl G. Distal pancreatectomy: incidence of postoperative diabetes. J Gastrointest Surg. 2008 Sep;12(9):1548-53. doi: 10.1007/s11605-008-0560-5. Epub 2008 Jun 10. PMID 18543045
- [Background] You DD, Choi SH, Choi DW, Heo JS, Ho CY, Kim WS. Long-term effects of pancreaticoduodenectomy on glucose metabolism. ANZ J Surg. 2012 Jun;82(6):447-51. doi: 10.1111/j.1445-2197.2012.06080.x. Epub 2012 May 9. PMID 22571457
- [Derived] Dai M, Xing C, Shi N, Wang S, Wu G, Liao Q, Zhang T, Chen G, Wu W, Guo J, Liu Z. Risk factors for new-onset diabetes mellitus after distal pancreatectomy. BMJ Open Diabetes Res Care. 2020 Oct;8(2):e001778. doi: 10.1136/bmjdrc-2020-001778. PMID 33122295